CLINICAL TRIAL: NCT03387852
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, 12-week Proof-of-Concept (PoC) Study to Assess the Efficacy, Safety, and Tolerability of SAR440340 and the Coadministration of SAR440340 and Dupilumab in Patients With Moderate-to-Severe Asthma Who Are Not Well Controlled on Inhaled Corticosteroid (ICS) Plus Long-acting β2 Adrenergic Agonist (LABA) Therapy
Brief Title: Evaluation of SAR440340 and as Combination Therapy With Dupilumab in Moderate-to-Severe Asthma Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACT15102; 2017-003289-29 (EudraCT Number); U1111-1194-2185 (Other: UTN)
Record Dates: First submitted 2017-12-15; First posted 2018-01-02 (Actual); Results first posted 2022-03-29 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — itepekimab; dupilumab; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- SAR440340 (Experimental): Participants received 2 injections of SAR440340 300 milligram (mg) along with 1 injection of dupilumab placebo, subcutaneous (SC) once every 2 weeks (Q2W) for 12 weeks.
  Interventions: Drug: SAR440340; Drug: Fluticasone or Fluticasone/salmeterol combination; Drug: Placebo for dupilumab
- Dupilumab (Active Comparator): Participants received 1 injection of dupilumab 300 mg along with 2 injections of SAR440340 placebo, SC Q2W for 12 weeks.
  Interventions: Drug: Dupilumab; Drug: Fluticasone or Fluticasone/salmeterol combination; Drug: Placebo for SAR440340
- SAR440340 + Dupilumab (Experimental): Participants received 2 injections of SAR440340 300 mg along with 1 injection of dupilumab 300 mg, SC Q2W for 12 weeks.
  Interventions: Drug: SAR440340; Drug: Dupilumab; Drug: Fluticasone or Fluticasone/salmeterol combination
- Placebo (Placebo Comparator): Participants received 2 SC injections of SAR440340 placebo along with 1 SC injection of dupilumab placebo Q2W for 12 weeks.
  Interventions: Drug: Fluticasone or Fluticasone/salmeterol combination; Drug: Placebo for SAR440340; Drug: Placebo for dupilumab

INTERVENTIONS:
Drug: SAR440340 — Pharmaceutical form: Solution for Injection, Route of administration: SC
  Other Names: REGN3500
  Arms: SAR440340; SAR440340 + Dupilumab
Drug: Dupilumab — Pharmaceutical form: Solution for Injection, Route of administration: SC
  Other Names: SAR231893 (REGN668)
  Arms: Dupilumab; SAR440340 + Dupilumab
Drug: Fluticasone or Fluticasone/salmeterol combination — Pharmaceutical form: Aerosol, dry powder, Route of administration: Inhaled
Drug: Placebo for SAR440340 — Pharmaceutical form: Solution for Injection, Route of administration: SC
  Arms: Dupilumab; Placebo
Drug: Placebo for dupilumab — Pharmaceutical form: Solution for Injection, Route of administration: SC
  Arms: Placebo; SAR440340

SUMMARY:
Primary Objective:

To evaluate the effects of SAR440340 with or without dupilumab, compared to placebo, on reducing the incidence of "loss of asthma control" (LOAC) events.

Secondary Objectives:

To evaluate the effects of SAR440340/REGN3500 and coadministration of SAR440340 and dupilumab, compared with placebo, on forced expiratory volume in 1 second (FEV1).

To evaluate the effects of coadministration of SAR440340 and dupilumab, compared with SAR440340 and compared with dupilumab, on FEV1.

To assess safety and tolerability of SAR440340 alone and in coadministration with dupilumab.

DETAILED DESCRIPTION:
The total duration of the study (per participant) was approximately 36 weeks, including 4 weeks screening, 12 weeks treatment, and 20 weeks post-treatment.

ELIGIBILITY:
Inclusion criteria :

* Adult participants with a physician diagnosis of asthma for at least 12 months based on the Global Initiative for Asthma (GINA) 2017 Guidelines.
* Participants with existing treatment with medium to high dose ICS (greater than or equal to [>=] 250 microgram (mcg) of fluticasone propionate twice a day (BID) or equipotent ICS daily dosage to a maximum of 2000 mcg/day of fluticasone propionate or clinically comparable) in combination with a LABA as second controller for at least 3 months with a stable dose >=1 month prior to Visit 1.
* Participants with pre-bronchodilator FEV1 greater than (>) 40 percent (%) of predicted normal at Visit 1/Screening. Pre-bronchodilator FEV1 >=50% but less than or equal to (<=) 85% of predicted normal at Visit 2/Baseline.
* Participants with reversibility of at least 12% and 200 milliliters (mL) in FEV1 after administration of 2 to 4 puffs (200-400 microgram [µg]) of albuterol/salbutamol or levalbuterol/levosalbutamol during screening or documented history of a reversibility test that meets this criteria within 12 months prior to Visit 1 or documented positive response to methacholine challenge (a decrease in FEV by 20% [PC20] of less than [<] 8 milligram per milliliter [mg/mL]) within 12 months prior to Visit 1/Screening is considered acceptable to meet this inclusion criterion.
* Participants had experienced, within 1 year prior to Visit 1, any of the following events at least once:
* Treatment with a systemic steroid (oral or parenteral) for worsening asthma.
* Hospitalization or emergency medical care visit for worsening asthma.
* Signed written informed consent.

Exclusion criteria:

* Participants <18 years or >70 years of age (i.e., have reached the age of 71 at the screening visit).
* Participants with body mass index (BMI) <16.
* Chronic lung disease (for example, chronic obstructive pulmonary disease [COPD], or idiopathic pulmonary fibrosis [IPF]), which might impair lung function.
* History of life threatening asthma (i.e., severe exacerbation that required intubation).
* Co-morbid disease that might interfere with the evaluation of investigational medicinal product (IMP).
* Participants with any of the following events within the 4 weeks prior to their Screening Visit 1:
* Treatment with 1 or more systemic (oral and/or parenteral) steroid bursts for worsening asthma;
* Hospitalization or emergency medical care visit for worsening asthma.
* Asthma Control Questionnaire 5-question version (ACQ-5) score <1.25 or >3.0 at Visit 2/randomization. During the screening period, an ACQ-5 of up to <=4 was acceptable.
* Anti-immunoglobulin E (IgE) therapy (e.g., omalizumab [Xolair®]) within 130 days prior to Visit 1 or any other biologic therapy (including anti interleukin-5 [anti-IL5] monoclonal antibodies [mAb]) or systemic immunosuppressant (e.g., methotrexate) to treat inflammatory disease or autoimmune disease (e.g., rheumatoid arthritis, inflammatory bowel disease, primary biliary cirrhosis, systemic lupus erythematosus, multiple sclerosis, etc.) and other diseases, within 2 months or 5 half-lives prior to Visit 1, whichever was longer.
* Participants with a history of a systemic hypersensitivity reaction to a biologic drug.
* Participants on or initiation of bronchial thermoplasty within 2 years prior to Visit 1 or plan to begin therapy during the screening period or the randomized treatment period.
* Current smoker or cessation of smoking within the 6 months prior to Visit 1.
* Previous smoker with a smoking history >10 pack-years.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2019-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (71):
- United States (18):
  - Investigational Site Number 8400026, Birmingham, Alabama
  - Investigational Site Number 8400004, Long Beach, California
  - Investigational Site Number 8400020, Los Angeles, California
  - Investigational Site Number 8400001, Rolling Hills Estates, California
  - Investigational Site Number 8400013, San Jose, California
  - Investigational Site Number 8400009, Stockton, California
  - Investigational Site Number 8400016, Colorado Springs, Colorado
  - Investigational Site Number 8400021, Ann Arbor, Michigan
  - Investigational Site Number 8400022, Minneapolis, Minnesota
  - Investigational Site Number 8400007, Papillion, Nebraska
  - Investigational Site Number 8400025, Edmond, Oklahoma
  - Investigational Site Number 8400011, Medford, Oregon
  - Investigational Site Number 8400024, Portland, Oregon
  - Investigational Site Number 8400010, Dallas, Texas
  - Investigational Site Number 8400023, Dallas, Texas
  - Investigational Site Number 8400006, Plano, Texas
  - Investigational Site Number 8400008, Murray, Utah
  - Investigational Site Number 8400014, Milwaukee, Wisconsin
- Argentina (5):
  - Investigational Site Number 0320001, Buenos Aires
  - Investigational Site Number 0320003, Caba
  - Investigational Site Number 0320002, Caba
  - Investigational Site Number 0320004, Caba
  - Investigational Site Number 0320005, Mendoza
- Chile (8):
  - Investigational Site Number 1520002, Quillota
  - Investigational Site Number 1520001, Santiago
  - Investigational Site Number 1520009, Santiago
  - Investigational Site Number 1520008, Santiago
  - Investigational Site Number 1520007, Santiago
  - Investigational Site Number 1520004, Santiago
  - Investigational Site Number 1520005, Talca
  - Investigational Site Number 1520003, Viña del Mar
- Mexico (6):
  - Investigational Site Number 4840005, Chihuahua City
  - Investigational Site Number 4840004, Durango
  - Investigational Site Number 4840002, Guadalajara
  - Investigational Site Number 4840006, Monterrey
  - Investigational Site Number 4840001, Monterrey
  - Investigational Site Number 4840003, Veracruz
- Poland (7):
  - Investigational Site Number 6160001, Bialystok
  - Investigational Site Number 6160008, Bialystok
  - Investigational Site Number 6160005, Bydgoszcz
  - Investigational Site Number 6160007, Krakow
  - Investigational Site Number 6160002, Poznan
  - Investigational Site Number 6160006, Poznan
  - Investigational Site Number 6160003, Żnin
- Russia (9):
  - Investigational Site Number 6430003, Moscow
  - Investigational Site Number 6430001, Moscow
  - Investigational Site Number 6430005, Moscow
  - Investigational Site Number 6430008, Ryazan
  - Investigational Site Number 6430007, Saint Petersburg
  - Investigational Site Number 6430010, Saint Petersburg
  - Investigational Site Number 6430006, Saint Petersburg
  - Investigational Site Number 6430009, Stavropol
  - Investigational Site Number 6430004, Ulyanovsk
- Turkey (Türkiye) (8):
  - Investigational Site Number 7920004, Ankara
  - Investigational Site Number 7920003, Bursa
  - Investigational Site Number 7920001, Istanbul
  - Investigational Site Number 7920006, Izmir
  - Investigational Site Number 7920007, Izmir
  - Investigational Site Number 7920008, Kırıkkale
  - Investigational Site Number 7920002, Mersin
  - Investigational Site Number 7920009, Rize
- Ukraine (10):
  - Investigational Site Number 8040008, Chernivtsi
  - Investigational Site Number 8040012, Ivano-Frankivsk
  - Investigational Site Number 8040002, Kharkiv
  - Investigational Site Number 8040009, Kharkiv
  - Investigational Site Number 8040011, Kharkiv
  - Investigational Site Number 8040007, Kyiv
  - Investigational Site Number 8040001, Kyiv
  - Investigational Site Number 8040006, Odesa
  - Investigational Site Number 8040003, Ternopil
  - Investigational Site Number 8040005, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Yin Z, Zhou Y, Turnquist HR, Liu Q. Neuro-epithelial-ILC2 crosstalk in barrier tissues. Trends Immunol. 2022 Nov;43(11):901-916. doi: 10.1016/j.it.2022.09.006. Epub 2022 Oct 14. PMID 36253275
- [Derived] Wechsler ME, Ruddy MK, Pavord ID, Israel E, Rabe KF, Ford LB, Maspero JF, Abdulai RM, Hu CC, Martincova R, Jessel A, Nivens MC, Amin N, Weinreich DM, Yancopoulos GD, Goulaouic H. Efficacy and Safety of Itepekimab in Patients with Moderate-to-Severe Asthma. N Engl J Med. 2021 Oct 28;385(18):1656-1668. doi: 10.1056/NEJMoa2024257. PMID 34706171

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 12-March-2018 to 7-August-2019. Participants were screened at 70 centers across 8 countries, out of which 68 centers randomized at least 1 participant.
Pre-assignment Details: A total of 499 participants were screened, out of which 296 participants were enrolled and randomized to 1 of the 4 treatment groups.
Groups:
- Placebo: Participants received 2 subcutaneous (SC) injections of SAR440340 placebo along with 1 SC injection of dupilumab placebo once every 2 weeks (Q2W) for 12 weeks.
- SAR440340 300 mg: Participants received 2 injections of SAR440340 300 milligram (mg) along with 1 injection of dupilumab placebo, SC Q2W for 12 weeks.
- Dupilumab 300 mg: Participants received 1 injection of dupilumab 300 mg along with 2 injections of SAR440340 placebo, SC Q2W for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | SAR440340 300 mg | SAR440340 + Dupilumab | Dupilumab 300 mg
Started (Randomized) | 74 | 73 | 74 | 75
Treated | 74 | 73 | 74 | 74
Completed | 41 | 55 | 47 | 56
Not Completed | 33 | 18 | 27 | 19
Not completed — Adverse event (AE) | 3 | 0 | 2 | 0
Not completed — Loss of asthma control (LOAC) | 28 | 16 | 20 | 14
Not completed — Withdrawal by participant | 1 | 1 | 3 | 2
Not completed — Other- Unspecified | 1 | 1 | 2 | 1
Not completed — Poor compliance to protocol | 0 | 0 | 0 | 1
Not completed — Randomized and not treated | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on randomized population that included any participant who had signed informed consent and had been allocated to a randomized treatment regardless of whether the treatment kit was used.
Groups:
- SAR440340 300 mg: Participants received 2 injections of SAR440340 300 mg along with 1 injection of dupilumab placebo, SC Q2W for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | SAR440340 300 mg | SAR440340 + Dupilumab | Dupilumab 300 mg | Total
Number analyzed (Participants) | 74 | 73 | 74 | 75 | 296
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.0 (11.4) | 49.0 (13.9) | 49.1 (12.0) | 51.3 (12.7) | 49.1 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 50 | 51 | 41 | 189
  Male | 27 | 23 | 23 | 34 | 107
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 1 | 1 | 4
  Asian | 0 | 2 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 2 | 0 | 6
  White | 71 | 68 | 69 | 73 | 281
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Loss of Asthma Control
Description: An LOAC event during the 12-week treatment period was a deterioration of asthma defined as any of the following: a) 30 percent (%) or greater reduction from baseline in morning peak expiratory flow (PEF) on 2 consecutive days; b) greater than or equal to (>=) 6 additional reliever puffs of salbutamol/albuterol or levosalbutamol/levalbuterol in a 24-hour period (compared to baseline) on 2 consecutive days; c) increase in inhaled corticosteroid (ICS) >=4 times the last prescribed ICS dose (or >=50% of the prescribed ICS dose at Baseline if background therapy withdrawal completed); d) required use of systemic (oral and/or parenteral) steroid treatment; e) required hospitalization or emergency room visit.
Time Frame: From Baseline up to Week 12
Population: The analysis was performed on modified intent-to-treat (mITT) population that included all randomized participants who have received at least 1 dose of investigational medicinal product (IMP) analyzed according to the treatment group allocated by randomization.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Participants received 2 SC injections of placebo matching to SAR440340 along with 1 SC injection of placebo matching to dupilumab once Q2W for 12 weeks.
- SAR440340 300 mg: Participants received 2 injections of SAR440340 300 mg along with 1 injection of placebo matching to dupilumab, SC Q2W for 12 weeks.
- Dupilumab 300 mg: Participants received 1 injection of dupilumab 300 mg along with 2 injections of placebo matched to SAR440340, SC Q2W for 12 weeks.
Arm/Group | Placebo | SAR440340 300 mg | SAR440340 + Dupilumab | Dupilumab 300 mg
Number analyzed (Participants) | 74 | 73 | 74 | 74
percentage of participants | 40.5 | 21.9 | 27.0 | 18.9
Statistical Analysis 1: Comparison: Placebo vs SAR440340 300 mg; Odds ratio, 95% confidence interval (CI), and p-value derived from logistic regression with treatment, baseline eosinophil strata, region, background ICS dose level at randomization and number of exacerbation events (defined as required use of systemic [oral and/or parenteral] steroid treatment, or required hospitalization or emergency room visit) within 1 year prior to screening; Test type: Superiority; p = 0.0214, Regression, Logistic; Odds ratio = 0.423, 95% CI 2-sided [0.203 to 0.88] — SAR440340 300 mg vs. Placebo
Statistical Analysis 2: Comparison: Placebo vs SAR440340 + Dupilumab; Odds ratio, 95% CI, and p-value derived from logistic regression with treatment, baseline eosinophil strata, region, background ICS dose level at randomization and number of exacerbation events (defined as required use of systemic [oral and/or parenteral] steroid treatment, or required hospitalization or emergency room visit) within 1 year prior to screening; Test type: Superiority; p = 0.0709, Regression, Logistic; Odds ratio = 0.520, 95% CI 2-sided [0.256 to 1.057] — SAR440340 + Dupilumab vs. Placebo

2. Secondary Outcome: Change From Baseline at Week 12 in Pre-bronchodilator Forced Expiratory Volume in 1 Second (FEV1)
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by spirometer. Pre-bronchodilator FEV1 refers to the spirometry performed after a wash period of bronchodilators (i.e., not earlier than 6 hours) after the last dose of albuterol/salbutamol or levalbuterol/levosalbutamol from a primed meter dose inhaler and withholding the last dose of long-acting β2 adrenergic agonist (LABA) for at least 12 hours, and prior to administration of study drug.
Time Frame: Baseline, Week 12
Population: Analysis was performed on mITT population. Here, "Overall number of participants analyzed" signifies participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: liters
Groups:
- Placebo: Participants received 2 SC injections of placebo matching to SAR440340 along with 1 SC injection of placebo matching to dupilumab Q2W for 12 weeks.
Arm/Group | Placebo | SAR440340 300 mg | SAR440340 + Dupilumab | Dupilumab 300 mg
Number analyzed (Participants) | 41 | 58 | 49 | 56
liters | 0.06 (0.35) | 0.11 (0.34) | 0.06 (0.37) | 0.14 (0.43)

3. Secondary Outcome: Change From Baseline at Week 12 in Post-bronchodilator Forced Expiratory Volume in 1 Second
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by spirometer. Post-bronchodilator FEV1 refers to the spirometry performed within 30 minutes after administration of bronchodilator.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | SAR440340 300 mg | SAR440340 + Dupilumab | Dupilumab 300 mg
Number analyzed (Participants) | 42 | 58 | 51 | 57
liters | -0.02 (0.27) | -0.00 (0.33) | 0.06 (0.41) | 0.09 (0.42)

ADVERSE EVENTS:
Time Frame: From first administration of IMP up to the final visit (Week 32) regardless of seriousness or relationship to IMP
Description: Analysis was performed on safety population that included all enrolled participants who had received at least 1 dose of study drug, analyzed as per actual treatment received.
Groups:
- SAR440340 300mg: Participants received 2 injections of SAR440340 300 mg along with 1 injection of dupilumab placebo, SC Q2W for 12 weeks.
- Dupilumab 300mg: Participants received 1 injection of dupilumab 300 mg along with 2 injections of SAR440340 placebo, SC Q2W for 12 weeks.
Arm/Group | Placebo | SAR440340 300mg | SAR440340 + Dupilumab | Dupilumab 300mg
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/73 | 0/74 | 1/74
Serious Adverse Events (participants affected / at risk) | 3/74 | 3/73 | 2/74 | 3/74
Other Adverse Events (participants affected / at risk) | 31/74 | 29/73 | 26/74 | 28/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=74) | SAR440340 300mg (N=73) | SAR440340 + Dupilumab (N=74) | Dupilumab 300mg (N=74)
Aortic Valve Incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess Jaw (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis Acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alcohol Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic Aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=74) | SAR440340 300mg (N=73) | SAR440340 + Dupilumab (N=74) | Dupilumab 300mg (N=74)
Nausea (Gastrointestinal disorders) | 2 (4) | 4 (4) | 2 (2) | 1 (1)
Injection Site Reaction (General disorders) | 4 (6) | 1 (1) | 5 (16) | 4 (4)
Nasopharyngitis (Infections and infestations) | 9 (10) | 13 (15) | 8 (8) | 9 (11)
Upper Respiratory Tract Infection Bacterial (Infections and infestations) | 2 (2) | 1 (1) | 4 (4) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 2 (3) | 1 (1) | 5 (7) | 3 (3)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 5 (6) | 3 (3) | 5 (7) | 2 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 7 (7) | 6 (7) | 5 (9) | 10 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 0 (0) | 1 (1)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 0 (0) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2018-09-06): https://cdn.clinicaltrials.gov/large-docs/52/NCT03387852/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-28): https://cdn.clinicaltrials.gov/large-docs/52/NCT03387852/SAP_001.pdf